CLINICAL TRIAL: NCT01136551
Title: An Open-label, Three-period, Crossover Study in Healthy Volunteers to Evaluate the Relative Bioavailability of Two Different Release Rate Controlled Release Formulations of Huperzine A (0.4mg)Compared to the Equivalent Dose of an Immediate Release Formulation.
Brief Title: Comparative Bioavailability Study of an Immediate Release and Controlled Release Oral Formulations of Huperzine A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Eliad Davidson, MD, School of pharmacy, Hebrew University of Jerusalem
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUPA - CR- HMO-CTIL; HUPA-HU-1 (Registry Identifier: Haddasah University Hospital)
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-05

CONDITIONS: Healthy; Bioavailability
Keywords: Pharmacokinetic profile of controlled release formulation of Huperzine A; Bioequivalence of Huperzine A IR formulation and CR formulation
MeSH Terms: interventions — huperzine A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IR formulation (Active Comparator): Healthy volunteers will receive imediate release formulation of Huperzine A (0.4mg)
  Interventions: Drug: Huperzine A
- CR 1 (Experimental): CR formulation
  Healthy volunteers will receive controlled release formulation 1 of Huperzine A (0.4mg)
  Interventions: Drug: Huperzine A
- CR 2 (Experimental): CR formulation
  Same volunteers will receive controlled release formulation 2 of Huperzine A (0.4mg)
  Interventions: Drug: Huperzine A

INTERVENTIONS:
Drug: Huperzine A — Each volunteer will receive single dose of three different formulations of Huperzine A. One immediate release formulation of 0.4mg and two different controlled release formulations at same dose. Between the study phases will be a washout period of at least 21 days.

SUMMARY:
The purpose of this study is to develop oral controlled release formulation of Huperzine A that will provide optimal pharmacokinetic profile of the drug enhancing safety and compliance, as possible cure to neurodegenerative disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males between the age of 18 and 35, inclusive (ASA = 1)
2. Body weight > 50 kg
3. Subject has a BMI less than 27 and more than 20
4. Participants should be able to ingest oral medication
5. The ability to understand and sign a written informed consent form, prior to participation and the willingness to comply with all study requirements

Exclusion Criteria:

1. History of drug sensitivity or drug allergy
2. History of sensitivity to eggs
3. Subject has a BMI less than 20 and more than 27
4. Previous participation in an investigational trial involving administration of any investigational compound within 1 month prior to the current study
5. History of alcoholism or drug addiction
6. Any medication taken including over-the-counter medications and herbal products within 14 days of commencing study drug dosing with the exception of vitamins and/or paracetamol. When a concomitant medication is necessary, this will be reviewed by the investigator and if not contraindicated, may be continued at the same dose and frequency during the study period
7. History of clinically important illness (ASA>1); Disorders or conditions that could affect the absorption, distribution, metabolism and/or excretion of drugs (e.g. malabsorption, edema, renal or hepatic insufficiency)
8. Inability to relate to and/or cooperate with the investigators
9. Blood loss or donation greater than 200ml in the 3 months prior to the trial
10. Exhausting physical exercise during the previous 48 hours to drug administration
11. Subjects who have smoked or used nicotine-containing products within 6 months prior to study entry

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-01 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of Huperzine A different formulations | Blood samples will be taken for 36 hours after Huperzine A administration
  Pharmacokinetic parameters: C max, T max, AUC, t1/2

SECONDARY OUTCOMES:
Laboratory testing of peripheral AchE inhibition by Huperzine A. Evaluation of adverse events. Laboratory testing of peripheral AchE inhibition by Huperzine A. Evaluation of adverse events. | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Friedman, Proffesor, Principal Investigator — Institute for Drug Research, Hebrew University of Jerusalem, Israel
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel